CLINICAL TRIAL: NCT00896792
Title: The Pilot Palliative ARNP (Advanced Registered Nurse Practitioner) Liaison Program (The PAL Program): Improving Communication Between Patients, Oncologists, and Hospice, Promoting Timely Hospice Referrals and Bringing Education and Research Efforts to Hospice and Palliative Care
Brief Title: Nurse Practitioner Hospice Program for Patients With Terminal Metastatic Cancer and Their Families or Caregivers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: CDR0000615562; P30CA015083 (NIH); MC0892 (Other: Mayo Clinic Cancer Center); 08-002293 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Hematopoietic/Lymphoid Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; hematopoietic/lymphoid cancer
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Counseling; Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: counseling intervention
Other: questionnaire administration
Other: survey administration
Procedure: end-of-life treatment/management
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Gathering information about patients with terminal metastatic cancer may help doctors learn more about the effectiveness of a nurse practitioner hospice program. It is not yet known whether a nurse practitioner program helps increase patients' length of stay in hospice.

PURPOSE: This randomized research study is evaluating a nurse practitioner hospice program for patients with terminal metastatic cancer and their families or caregivers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of the palliative advanced registered nurse practitioner liaison program (PAL) on length of patient's enrollment in hospice care.

Secondary

* To evaluate the impact of the PAL program on patient's knowledge about hospice services.
* To evaluate the impact of the PAL program on patient and family or caregiver's psychological stress during palliative treatments.

OUTLINE: Patients are randomized to 1 of 2 arms.

* Arm I (advanced registered nurse practitioner [ARNP] intervention): Patients and their families or caregiver receive information from an ARNP about terminal cancer, resources available for supportive care, and the benefits of palliative care. After transition to hospice, patients receive pain and palliative medicine, psychology, social services, chaplaincy, and patient support group intervention arranged by the ARNP. Patients complete the Patient Questionnaire about overall quality of life and mental, emotional, and physical well being at baseline and at 3 weeks after intervention or at time of enrollment in hospice. Patients and their families or caregivers are contacted by the ARNP weekly.
* Arm II (no ARNP intervention): Patients and their families or caregivers complete the same Patient Questionnaire, administered by a clinical research assistant (CRA), as in Arm I. Patients and their families or caregivers receive no ARNP intervention. After transition to hospice, patients receive routine hospice care.

Patients participate in this study for a duration of 21 days while in hospice care. At the completion of the study, patients in both arms complete questionnaires about pain management, social, emotional, and spiritual and mental well-being. Patients' families or caregivers complete the Caregiver Questionnaire and the Hospice Family Satisfaction Survey 3 weeks after patient's death.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of terminal metastatic cancer
* Patient at Mayo Clinic in Jacksonville, Florida
* Strong candidate for hospice care
* Entering or planning to enter Community Hospice of Northeast Florida

  * Willing to undergo visits by an Advanced Registered Nurse Practitioner (ARNP) after hospice enrollment

PATIENT CHARACTERISTICS:

* Willing to participate in 2 palliative care consultations with an ARNP prior to hospice enrollment
* Life expectancy < 12 months
* Able to complete questionnaires with or without assistance
* Has a primary caregiver with an identified relationship to the patient

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10-10 (Actual); Primary Completion 2009-11-20 (Actual); Study Completion 2015-03-17 (Actual)

PRIMARY OUTCOMES:
Increased length of enrollment time in hospice care

SECONDARY OUTCOMES:
Effects of incorporating a palliative care advanced registered nurse practitioner liaison program in the late-stage cancer care process
Increased knowledge of hospice services as assessed by a knowledge survey
Patient and family or caregiver psychological stress, as measured by the functional assessment of cancer therapy general (FACT-G) survey

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Colon-Otero, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic in Jacksonville, Jacksonville, Florida, United States